CLINICAL TRIAL: NCT01582568
Title: EUS Evaluation of Perianal and Peri-rectal Fistulizing Crohn's Disease With CERTOLIZUMAB Treatment
Acronym: EUS
Status: Terminated | Type: Observational
Why Stopped: Not enough subjects to reach accrual goals.
Sponsor: Baylor College of Medicine (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, Joseph Sellin, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-26958
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Crohns Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Certolizumab: Subjects will take the study drug certolizumab for 8 weeks. They will undergo a endoscopy before study drug and then again after study is complete. The study doctor will be looking for complete closure of the peri-anal fistula identified at visit 1 after the use of certolizumab based on and endoscopic ultrasound (EUS).
  Interventions: Drug: Certolizumab

INTERVENTIONS:
Drug: Certolizumab — Certolizumab 200mg-400mg subcutaneous every 2 weeks for 8 weeks.
  Other Names: Cimzia

SUMMARY:
The primary objective of this study is to assess perianal and perirectal fistula healing (complete closure) based on endoscopic ultrasound (EUS) evaluation at 3 months and by PDAI (Pouchitis Disease Activity Index) and Fistula Drainage assessment by 6 months, showing no fistula (new or recurrence) in treatment of Crohn's' disease patient with Certolizumab (Cimzia).

DETAILED DESCRIPTION:
Peri-anal ( located around the anus, the opening of the rectum to the outside of the body) fistulae are a major complication of Crohn's disease and occur in almost 30% of patients. Patients with perianal fistulae suffer from severe pain, perianal drainage, and have significant impairment of quality of life. Initial studies of Infliximab and Adalimumab in patients with CD have shown perianal fistula healing with these medications. Infliximab and Adalimumab are medications which reduce the effects of a substance in the body that can cause inflammation. They are also used to treat Crohn's disease after other drugs have been tried without successful treatment of symptoms. Although no studies have specifically evaluated Certolizumab (Cimzia) treatment in fistulizing Crohn's disease, there is evidence to its efficacy. Certolizumab reduces the effects of a substance in the body that can cause inflammation. Certolizumab is used to treat the symptoms of Crohn's disease after other drugs have been tried without successful treatment of symptoms. Studies with a small number of patients who use Cimzia did not show any significant effect on fistula closure. However, in a larger subgroup of patients with fistulae in PRECiSE 2 43.3% of those who received 3 induction injections of certolizumab followed by placebo, and 53.6% of those on certolizumab 400mg continuous treatment had fistula closure defined as no drainage on gentle compression of at least 50% of open fistulae at any 2 consecutive visits, at least 3 weeks apart. Perianal disease activity is usually monitored clinically. In clinical studies, two evaluation methods have been used in attempts to unify the definition of perianal disease activity. One method is the perianal Crohn's disease activity index (PDAI) which involves questions regarding discharge, pain/ restriction of activities, restriction of sexual activity, type of perianal disease, degree of induration (with scores >/=5 indicating active disease, with decrease in PDAI of 2 or more points indicates improvement, and consider 0 as healed. PDAI scale (Pouchitis Disease Activity Index). This scale analyzes and summarizes different criteria: clinical, endoscopic and histological. Among clinical symptoms, an important factor is the number of stools exceeding the post-operative average, bleeding, re-occuring stomachaches, as well as body temperature above 37.8°C or 100°F. "Pouchitis" is a term to describe inflammatory changes in the pouch created from the lower part of the ileum. The patients suffer from high body temperature, stomachaches and watery stools with small amounts of mucus, blood and soiling. An exam based technique, used in the Precise trials is the Fistula Drainage Assessment indicating improvement or remission with closure of individual fistulae defined as no fistula drainage despite gentle finger compression, improvement defined as a decrease from baseline in the number of open draining fistulae of greater than or equal to 50 percent for at least 2 consecutive visits (i.e. at least 4 weeks), and remission defined as closure of all fistulae that were draining at baseline for at least 2 consecutive visits (i.e., at least 4 weeks). However both have not been validated, and the response levels are usually evaluated several months into treatment. If another method could provide early assessment / predictors of healing, it could make the decision for the treatment of the gastroenterologist as well as the patient, easier to determine if they should continue the biologic or stop. Studies have evaluated the use of endoscopic ultrasound (EUS) to follow fistula assessment and healing, but none have specifically assessed this in response to certolizumab treatment. EUS is increasingly used and has been found to be equally accurate in the evaluation of perianal fistulae compared to MRI of the pelvis. An accurate assessment and classification of fistulae can facilitate further management including surgical planning, further medical treatment, or a combination of both. EUS can evaluate for fistulae as well as abscesses and the relation to the anatomic landmarks of the rectum including the sphincter muscles as well as adjacent organs such as vagina and the bladder. EUS has the advantage of being more convenient for the patient than an MRI. An MRI can take a long duration, can cause anxiety in those that are claustrophobic, and is expensive. EUS is usually performed with sedation and by the treating physician allowing a more personal evaluation of the fistula anatomy and correlation of endoscopic mucosal findings. Thus, we propose to evaluate the use of certolizumab in Crohn's disease patients with peri-anal and peri-rectal fistulae (an abnormal passage that leads from an abscess or hollow organ or part to the body surface or from one hollow organ or part to another) and to assess their response and healing (A perirectal abscess is a collection of pus in the deep tissues surrounding the anus. Perirectal and perianal abscesses are thought to develop from the glands surrounding the anus) based on EUS findings. This study can help provide recommendations on fistula classification of EUS and use this classification to provide EUS - based early predictors of response of treatment with certolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Conventional therapy here indicates non-biologic therapy. Study subjects would have failed conventional and standard regimens of treatment such as immunomodulators (azathioprine, 6-mercaptopurine, methotrexate) or mesalamines or corticosteroids. Certolizumab is actually an approved regimen of treatment for Crohn's disease as patients with perianal fistulas fall under those with moderately to severely active disease. It is not an off-label indication, therefore would not require an IND. The study goal is to look at EUS as a tool to determine how fistula healing occurs with the use of certolizumab which is one of the biologic therapies used to treat fistulizing Crohn's disease. Crohn's disease patients with peri-anal or peri-rectal fistulizing disease. Moderate to severe Crohn's disease patients between the ages of 18 and 70 years with active peri-anal or peri-rectal fistula.

Exclusion Criteria:

* Pre-existing fistula improving on current medical therapy. Contraindication to certolizumab use. Prior use of anti-TNF-alpha.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Crohn's disease patients with peri-anal or peri-rectal fistulizing disease. Moderate to severe Crohn's disease patients between the ages of 18 and 70 years with active peri-anal or peri-rectal fistula.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The response rate | 6 months
  The primary objective of this study is to assess perianal and perirectal fistula healing (complete closure) based on endoscopic ultrasound (EUS) evaluation at 3 months and by PDAI (Pouchitis Disease Activity Index) and Fistula Drainage assessment by 6 months, showing no fistula (new or recurrence) on treatment of Certolizumab (Cimzia) in Crohn's's disease patient s.

SECONDARY OUTCOMES:
Fistula healing based on EUS | 6 months
  The secondary objectives: 1. To define an Endoscopic Ultrasound (EUS)-based classification system which will compare and analyze perianal and perirectal fistulizing (abnormal opening between two hollow organs) in Crohn's disease. 2. To compare the EUS classification to PDAI and Fistula Drainage Assessment scores. 3. To determine EUS-based early predictors which can be summarized by the findings/results of the EUS procedure of fistula healing with Certolizumab (Cimzia) treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bincy P. Abraham, MD, MS, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No